CLINICAL TRIAL: NCT00700804
Title: Meat Protein and Calcium: Do They Interact Synergistically or Antagonistically?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: GFHNRC064; IRB-200307-010
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-05

CONDITIONS: Dietary Proteins
Keywords: Calcium retention; dietary protein; dietary calcium
MeSH Terms: interventions — Diet, High-Protein; Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Calcium Diet (Experimental)
  Interventions: Behavioral: High Protein Diet
- Low Calcium Diet (Experimental)
  Interventions: Behavioral: Low Protein Diet

INTERVENTIONS:
Behavioral: High Protein Diet — High and low protein diets with meat as a primary protein source, tested in a cross-over design for each arm
  Arms: High Calcium Diet
Behavioral: Low Protein Diet — High and low protein diets with meat as a primary protein source, tested in a cross-over design for each arm
  Arms: Low Calcium Diet

SUMMARY:
The primary objective is to determine whether meat interacts positively with calcium to improve calcium retention. The secondary objective is to determine whether any interaction between dietary protein and calcium affects biomarkers of bone metabolism.

DETAILED DESCRIPTION:
This study tests the effects of dietary protein and calcium on calcium retention and indices of bone metabolism. It is a controlled feeding trial with a randomized crossover design (2x2 Factorial), studying 34 healthy post-menopausal women. The women are blocked on Body Mass Index (weight in kilograms divided by height in meters squared)and randomly assigned to a high calcium (HC,1500 milligrams per day) or low calcium (LC, 600 milligrams per day) group, and consume both low protein (LP,10% protein) and high protein (HP, 20% protein) diets for 7 weeks each. There is a 3-week "washout" between dietary periods, during which the subjects consume self-selected diets. After 3 week equilibration to each diet, the 2-day rotating menu is extrinsically labeled with a Calcium-47 radiotracer and retention is monitored for 28 days by whole body scintillation counting. In addition to Calcium retention, other endpoints include urinary indices of acid excretion and urine serum indices of bone resorption.

ELIGIBILITY:
Inclusion Criteria:

* at least 3 years since last menses
* bone mineral density equal to or greater than 2.5 standard deviations from average bone mineral density for young adults,
* body mass index equal to or less than 35 kilograms/meter squared

Exclusion Criteria:

* taking prescription medication other than hormone replacement therapy

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-06; Primary Completion 2004-07 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet R Hunt, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- United States Department of Agriculture (USDA) Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Post menopausal women willing to eat controlled diet at United States Department of Agriculture (USDA) Grand Forks Human Nutrition Research Center for 14 weeks
Pre-assignment Details: Subjects were assigned to either the High or Low Calcium diets. The subjects then consumed the high and low protein diets in random order, i.e. half of the subjects consumed high protein, then low protein while the other half consumed low protein, then the high protein diet. Drop-outs were replaced.
Groups:
- High Calcium Diet: Women consumed diets containing 1500 milligrams of calcium daily
- Low Calcium Diet: Women consumed diets containing 600 milligrams of calcium daily
Period: Overall Study
Arm/Group | High Calcium Diet | Low Calcium Diet
Started | 17 | 17
Completed | 14 | 13
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Loose Stools | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Calcium Diet | Low Calcium Diet | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (5) | 58 (6) | 57 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Serum Insulin-like Growth Factor 1 (IGF-1)
Time Frame: 7 weeks
Measure: Geometric Mean (Standard Error); unit: nanomoles per liter (nmols/L)
Arm/Group | High Calcium Diet | Low Calcium Diet
Number analyzed (Participants) | 14 | 13
nanomoles per liter (nmols/L)
  High Protein Diet | 5.23 (0.12) | 5.07 (0.12)
  Low Protein Diet | 4.96 (0.12) | 4.87 (0.12)

2. Primary Outcome: Calcium Absorption
Description: Retention of Calcium-47 was monitored for 28 days by whole body scintillation counting. The percentage of Calcium-47 absorbed was estimated from the y-intercept of the linear portion of a semilogarithmic retention plot of percent Calcium-47 retained vs time
Time Frame: 17 weeks
Population: Only participants which completed both protein diet periods were included in the statistical analysis
Measure: Mean (Standard Deviation); unit: percentage of Calcium absorbed
Arm/Group | High Calcium Diet | Low Calcium Diet
Number analyzed (Participants) | 14 | 13
percentage of Calcium absorbed
  High Protein Diet | 18.1 (2.5) | 29.5 (2.5)
  Low Protein Diet | 18.0 (2.5) | 26 (2.5)
Statistical Analysis 1: Comparison: High Calcium Diet vs Low Calcium Diet; Test type: Superiority or Other; p = 0.05, Mixed Models Analysis; Effects of calcium (Ca), protein & their interaction were tested using repeated measures analysis of variance (subjects nested under High or Low Ca); Mean Difference (Final Values) = 9.7, Standard Deviation 2.5 — Reported analysis is the main effect of Calcium (High vs Low) from the Mixed Model Analysis which averages across the two levels of dietary protein. The main effect of protein and the calcium x protein interaction were not statistically significant

ADVERSE EVENTS:
Arm/Group | High Calcium Diet | Low Calcium Diet
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes